CLINICAL TRIAL: NCT03978663
Title: Evaluating the Use of Stereotactic Radiation Therapy Prior to Neoadjuvant Chemotherapy for High-risk Breast Carcinoma (a SIGNAL Series Clinical Trial): Three Fraction Radiation to Induce Immuno-Oncologic Response (TRIO Trial)
Brief Title: Three Fraction Radiation to Induce Immuno-Oncologic Response
Acronym: TRIO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 112626
Record Dates: First submitted 2019-06-01; First posted 2019-06-07 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: High-Risk Cancer; Locally Advanced Breast Cancer
Keywords: locally advanced breast cancer; immune priming; radiation therapy; neoadjuvant radiation; radiotherapy; immuno-oncology
MeSH Terms: interventions — Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant radiotherapy (Experimental): 3 doses of stereotactic radiotherapy administered prior to neoadjuvant chemotherapy in high-risk breast cancers.
  Interventions: Radiation: Neoadjuvant radiotherapy

INTERVENTIONS:
Radiation: Neoadjuvant radiotherapy — Neoadjuvant radiation therapy delivered to a portion of the index tumour for high-risk breast carcinoma for immune priming prior to neoadjuvant radiation

SUMMARY:
Patients with high risk breast cancers (any locally advanced breast cancer patient defined as Stages IIB-III [excluding inflammatory breast cancer] with stage IIA being eligible for triple negative and HER2-positive breast cancers) will receive neoadjuvant radiation to any portion of their tumour in three fractions in order to act as an immune primer. Radiation will be delivered to a portion of the tumour in three fractions. The patient will be positioned prone as per the SIGNAL 2.0 protocol. The patient will then go on to standard of care treatment (neoadjuvant chemotherapy and surgery) followed by whole-breast radiation as needed. Pathologic complete response will be the primary outcome. Immune markers will also be evaluated.

DETAILED DESCRIPTION:
Patients eligible for neoadjuvant chemotherapy for locally advanced stage III (non-inflammatory) breast cancer or stage IIb (triple negative or Her2+) breast cancers will be approached to participate in this single arm trial. Patients with staging investigations ruling out distant disease will be approached to participate and will undergo pre-treatment image guided core biopsy and blood samples for molecular correlative studies, followed by hypofractionated radiation (delivered prone) to entire tumor with dose constraints to skin, critical organs and contralateral breast, plus a 0.5 cm PTV. As much of the tumor that can receive planned dose of 8 Gy per fraction x 3 fractions every second day, with fall off dose to 4 Gy per fraction x 3 fractions for PTV margin. Two weeks following completion of radiation, patients will undergo a second image guided core needle biopsy of tumor and blood sample. They will then begin standard neoadjuvant chemotherapy (anthracycline and taxane based), followed by a third tissue biopsy under image guidance of any residual tumor and blood sample and then standard surgery (breast conserving or lumpectomy). This will be followed by standard whole breast radiation (50 Gy in 25 fractions). Herceptin therapy and hormonal therapy will be administered as per clinical standard when indicated. Primary outcome will be measured as pathological complete response to treatment, and secondary outcomes will include toxicity, immune markers (tumor infiltrating lymphocytes, PD-1 and PD-L1 up-regulation and changes to the circulating lymphocyte counts.

ELIGIBILITY:
Inclusion Criteria:

1. Any biopsy-proven locally advanced breast cancer patient defined as Stages IIB-III (excluding inflammatory breast cancer). Stage IIA is eligible for triple negative and HER2-positive breast cancers
2. Invasive mammary carcinoma of any subtype excluding lobular, sarcomatous, or metaplastic subtypes, or with lobular features
3. Plan to be treated with neoadjuvant chemotherapy
4. Able to fit in/have MRI
5. 18 years of age or older
6. Able to tolerate core needle biopsies
7. Able to provide informed consent
8. No evidence of metastatic disease

Exclusion Criteria:

1. Any serious medical comorbidities or other contraindications to radiotherapy, chemotherapy, or surgery
2. Prior treatment for current breast cancer
3. Previous radiation therapy to the same breast
4. Inflammatory breast carcinoma
5. Invasive lobular carcinoma or invasive mammary carcinoma with lobular, sarcomatous, or metaplastic subtypes, or with lobular features
6. Recurrent breast cancer
7. Bilateral breast cancer
8. Evidence of distant metastatic disease
9. Collagen vascular disease (particularly lupus, scleroderma, dermatomyositis, psoriatic arthritis)
10. Any other malignancy at any site (except non-melanomatous skin cancer) <5 years prior to study enrollment
11. Inability to lay prone with arms above the head for extended periods of time
12. Inability to fit in/have an MRI
13. Inability to tolerate core needle biopsies
14. Pregnant or lactating
15. Under 18 years of age
16. Inability or unwillingness to provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-09-02 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response | Measured at time of surgery, typically 6 months after enrollment in trial.
  Pathologic complete response rates after neoadjuvant radiotherapy and chemotherapy will be evaluated.

SECONDARY OUTCOMES:
Response rates in the primary post chemotherapy by imaging | Measured after neoadjuvant radiation and chemotherapy has been completed, prior to surgery, typically 6 months after enrollment in trial.
  Response rates in the primary post chemotherapy by MRI +/- PET scan compared to pre-neoadjuvant radiation imaging
Response rates in the axillary nodes post chemotherapy by imaging and pathology | Measured after neoadjuvant radiation and chemotherapy has been completed, prior to surgery (imaging) and at time of surgery, typically 6 months after enrollment in trial.
  Absence of any invasive breast cancer cells in any tissue at time of surgery
Immune priming | Measured 14-20 days after the last dose of neoadjuvant radiation, prior to the start of neoadjuvant chemotherapy.
  Immune priming as measured by amount of tumour infiltrating lymphocytes (CD8) into tumour specimen, as well as the expression of immune markers (PDL1, Fox3) and immune panel in blood (CD4, CD8, neutrophil, and macrophage counts). Angiogenesis will be examined using the CD31 or VEGF-a cell markers, proliferation will be examined using the Ki67 marker, hypoxia will be examined using the Carbonic Anhydrase 9 (CAH IX), or HIF1/HIF2 markers, apoptosis will be examined using the Caspase-3, or Tunnel markers, invasion will be analyzed using the vimentin, or SDF1-a markers.
Radiation toxicity | Measured at study enrollment, at first surgical follow-up post-surgery, 6 months post surgery, and 1 year post surgery.
  Toxicity to surrounding breast and skin tissue, defined by ≥ grade 2 fibrosis.
Surgical wound healing and the overall complication rate. | Measured at the first surgical follow-up post-surgery, 6 months post surgery, and 1 year post surgery.
  Percentage of patients experiencing wound infection that requires wound to be opened and/or packed.
Local recurrence rates | Disease status will be evaluated at routine patient follow-up appointments, including yearly mammography. Will be reported at year 3.
  Ipsilateral breast recurrence rate.
Ability of imaging to predict patient response to radiotherapy. | Pre-treatment imaging to be done after study enrollment (baseline) and 14-20 days after the last dose of neoadjuvant radiation has been delivered.
  Correlation between complete clinical response on imaging and pathological complete response.
Ability of imaging markers to predict response to radiotherapy | Pre-treatment imaging to be done after study enrollment (baseline measurements) and 14-20 days after the last dose of neoadjuvant radiation has been delivered.
  Ability of FDG uptake, choline levels, perfusion, and ADC obtained from post-radiotherapy imaging to predict tissue response to high dose radiotherapy.
Ability to predict pathological response to treatment based on tumour genetics | Tissue samples for analysis will be taken 14-20 days after completion of neoadjuvant radiation, prior to the start of neoadjuvant chemotherapy and will be compared with tissue taken prior to the start of neoadjuvant radiation.
  Ability to predict pathological response to treatment based on microarray analysis of tumor gene expression.

CONTACTS AND LOCATIONS:
Overall Officials: Muriel Brackstone, MD PhD, Principal Investigator — London Health Sciences Centre/Lawson Health Research Institute; Michael Lock, MD, Study Chair — London Health Sciences Centre/London Regional Cancer Program; Brian Yaremko, MD, Study Chair — London Health Sciences Centre/London Regional Cancer Program
Locations (1):
- London Regional Cancer Program, London, Ontario, Canada